CLINICAL TRIAL: NCT04885946
Title: Fecal Microbiota Transplantation for Early Clostridioides Difficile Infection
Acronym: EarlyFMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Christian Hvas (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Sponsor-Investigator, Christian Hvas, MD PhD Consultant, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1-10-72-254-20
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Clostridium Difficile Infection; Clostridioides Difficile Infection
Keywords: Fecal microbiota tranplantation, FMT, CDI
MeSH Terms: conditions — Clostridium Infections; Diabetes Insipidus, Neurogenic

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either vancomycin + 2 FMT or 2 placebo. An open-label arm exists for patients with fulminant CDI.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vancomycin 125 x 4 for 10 days + 2 Fecal Microbota Transplantation (Experimental): Patients are required to undergo full treatment with vancomycin and are randomized following completion to, in this arm, FMT.
  Interventions: Other: Fecal microbiota transplantion (FMT)
- Vancomycin 125 x 4 for 10 days + 2 Placebo (Placebo Comparator): Patients are required to undergo full treatment with vancomycin and are randomized following completion to, in this arm, placebo.
  Interventions: Other: Placebo
- Open-label for screened, but not randomized patients with fulminant CDI (Other): This arm exists for patients with fulminant CDI and for randomization to placebo may be considered unethical.
  Interventions: Other: Fecal microbiota transplantion (FMT)

INTERVENTIONS:
Other: Fecal microbiota transplantion (FMT) — Single donor, fecal microbiota transplantion (FMT) from healthy human donors.
  Arms: Open-label for screened, but not randomized patients with fulminant CDI; Vancomycin 125 x 4 for 10 days + 2 Fecal Microbota Transplantation
Other: Placebo — Food coloring, water, glycerol
  Arms: Vancomycin 125 x 4 for 10 days + 2 Placebo

SUMMARY:
Clostridioides difficile (CD) infection (CDI) is a global health threat with an urgent need for new treatment strategies. Faecal microbiota transplantation (FMT) is effective for recurrent Clostridioides difficile infection (CDI), and is currently recommended for multiple (three or more), recurrent CDI infections. The role of FMT earlier in the treatment hierarchy of CDI remains to be determined.

In this randomized, double-blinded, placebo-controlled clinical trial, we compare FMT with placebo following standard antibiotic treatment for first or second Clostridioides difficile infection.

DETAILED DESCRIPTION:
This is a parallel arm placebo-controlled clinical trial. We aim to include 84 adult patients with their first or second episode of Clostridioides difficile (formerly Clostridium difficile) infection. All patients receive vancomycin standard therapy. Patients are randomised in a 1:1 ratio to two treatments with capsules that contain either FMT+FMT or placebo+placebo. The primary outcome is absence of C difficile-associated disease 8 weeks after randomisation. Patients who have fulminant disease where it is deemed unethical to give placebo are offered open-label FMT. The primary outcome in patients with fulminant C difficile infection is 8 weeks mortality.

ELIGIBILITY:
Inclusion Criteria:

* 1. or 2. CDI (within a year) defined as: > 3 bowel movements of Bristol 6-7 per day and positive stool CD-test.
* Age 18 years or higher.

Exclusion Criteria:

* Pregnancy
* Does not speak or understand the Danish language
* Current antibiotic treatment other than vancomycin
* Current treatment with potential interations with vancomycin
* Allergy to vancomycin
* Previous anaphylactic reactions due to food allergies
* Continuous need for proton pump inhibitor
* Documented gastroparesis
* Fulminant CDI

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Resolution of CD-associated diarrhea (CDAD) week 8 | 8 weeks following treatment
  Measured as a combined clinical resolution or persistent diarrhea, but with negative CD test.
Mortality week 8 | 8 weeks following treatment
  In the open-label arm for patients who cannot be randomized due to ethical reasons, the primary outcome is mortality.

SECONDARY OUTCOMES:
Resolution of CD-associated diarrhea (CDAD) week 1 | 1 week following treatment
  Measured as a combined clinical resolution or persistent diarrhea, but with negative CD test.
Negative CD toxin-test week 1 | 1 week following treatment
  Faecal C difficile PCR test
Negative CD toxin-test week 8 | 8 weeks following treatment
  Faecal C difficile PCR test
Mortality week 8 | 8 weeks
  Date of death
Colectomy rate week 8 | 8 weeks
  Date of colectomy
Health-related quality of life | 8 weeks
  EDQ5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Hvas, PhD, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Data may be obtained in a anonymous form compliant with the General Data Protection Regulation (GDPR)

REFERENCES:
- [Derived] Baunwall SMD, Andreasen SE, Hansen MM, Kelsen J, Hoyer KL, Ragard N, Eriksen LL, Stoy S, Rubak T, Damsgaard EMS, Mikkelsen S, Erikstrup C, Dahlerup JF, Hvas CL. Faecal microbiota transplantation for first or second Clostridioides difficile infection (EarlyFMT): a randomised, double-blind, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2022 Dec;7(12):1083-1091. doi: 10.1016/S2468-1253(22)00276-X. Epub 2022 Sep 22. PMID 36152636